CLINICAL TRIAL: NCT01191983
Title: A Single Arm Open Label Multicenter Interventional Study to Assess the Efficacy, Safety, and Tolerability of Every 4 Weeks Administration of Subcutaneous C.E.R.A. for the Treatment of Chronic Renal Anemia in Diabetic Nephropathy With Chronic Kidney Disease Stages III-IV Not on Dialysis, Not Currently Treated With ESA.
Brief Title: A Study of Methoxy Polyethylene Glycol-Epoetin Beta (Mircera) for the Treatment of Chronic Renal Anemia in Participants With Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25276
Record Dates: First submitted 2010-08-16; First posted 2010-08-31 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methoxy polyethylene glycol-epoetin beta (Experimental): Participants will receive 1.2 mcg/kg methoxy polyethylene glycol-epoetin beta given in monthly doses at each visit. Dose will be measured on the basis of the participants Hb level during the study period. The dose administration will be the nearest possible dose using the prefilled syringes containing 50, 75 and 100 mcg/kg Q4W.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta [Mircera] — Starting dose of 1.2 mcg/kg, adjusted according to Hb values, administered by subcutaneous injection Q4W
  Other Names: Mircera, C.E.R.A

SUMMARY:
This single arm, open label study will assess the efficacy, safety and tolerability of methoxy polyethylene glycol-epoetin beta for the treatment of chronic renal anemia in participants with chronic kidney disease (CKD) secondary to diabetes. Participants who are not on dialysis and not currently treated with erythropoiesis stimulating agents (ESAs) will receive methoxy polyethylene glycol-epoetin beta subcutaneously every 4 weeks (Q4W). The starting dose of 1.2 microgram/kilogram (mcg/kg) methoxy polyethylene glycol-epoetin beta will be adjusted according to hemoglobin levels. Anticipated time on study treatment is 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic nephropathy
* Chronic renal anemia with stage III-IV CKD
* Not on dialysis and not expected to require dialysis within the next 6 months
* Not receiving any ESA in the 2 months prior to study
* Adequate iron status

Exclusion Criteria:

* Transfusion of red blood cells during the previous 2 months
* Known or clinical suspicion of pure red cell aplasia
* Hypersensitivity to recombinant human erythropoietin, polyethylene glycol or to any constituent of the study medication
* Haemoglobinopathy
* Significant acute or chronic bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-08-13 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Mean time taken to achieve target hemoglobin (Hb) levels range (10-12 g/dL) During Efficacy Evaluation Period (EEP) | EEP (Week 17 up to Week 24)
Change in Hb Concentration Between Baseline and EEP | Baseline (Week -2 up to Week 0); EEP (Week 17 up to Week 24)
Percentage of Participants Maintaining Hb Concentration Within the Target Range (10-12 g/dL) During EEP | EEP: (Week 17 up to Week 24)

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events | Baseline (Week -2 up to Week 0) to Week 28
Percentage of Participants With Red Blood Cell Transfusion During Treatment Period | Week 0 up to Week 24
Percentage of Participants with anti-epoetin antibodies | Baseline (Week-2 up to Week 0) up to Week 28
Short Form-36 Health Survey (SF-36) score | Week 0 to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- India (14):
  - Osmania General Hospital; Department of Nephrology, Hyderabad, Andhra Pradesh
  - Pushpawati Singhania Research Institute; Nephrology, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Vijayratna Diabetes Diagnosis & Treatment Center, Ahmedabad
  - M S Ramaiah Memorial Hospital, Bangalore
  - North Delhi Diabetes Centre, Delhi
  - MAX Balaji Hospital, Delhi
  - Dr.Modi's Clinic, Hyderabad
  - IPGMER & SSKM Hospital; Rheumatology and Clinical Immunology Centre, Kolkata
  - Apex Kidney Care Pvt. Ltd., Sushrut Hospital, Mumbai
  - Diab Care Centre, Mumbai
  - Sanjeevani Hospital, Mumbai
  - Sahyadri Speciality Hospital, Pune
  - Diabetes Care & Research Centre, Pune